CLINICAL TRIAL: NCT03800862
Title: The Role of Computed Tomography-Derived Fractional Flow Reserve (CT-FFR) and Myocardial Computed Tomographic Perfusion (CTP) in Patients Presenting With Chest Discomfort
Brief Title: The Evaluation of the Roles of New Cardiac Imaging in Patients With Chest Pain
Status: Terminated | Type: Observational
Why Stopped: PI departure from institution + Enrollment Challenges
Sponsor: Lancaster General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HEVA2018_RJ0002
Record Dates: First submitted 2018-12-17; First posted 2019-01-11 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Cardiology; Radiology; Stenoses
Keywords: Stenoses; Chest pain; Myocardial Infarction; Heart Attack; Radiology; Cardiac Imaging; Coronary artery disease
MeSH Terms: conditions — Constriction, Pathologic; Chest Pain; Myocardial Infarction; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- CTP and CT-FFR: This will be a prospective, observational study designed to include a convenience sample of all qualifying patients undergoing myocardial CTP and CT-FFR.
  The study will enroll patients who have chest discomfort and will require further evaluation for the presence of coronary artery disease. Patients in the study will include those who have had a clinically indicated CCTA for suspicion of coronary artery disease and are determined to have a coronary stenosis ≥50% and ≤99%. However, patients with Left main disease greater than 50% and occluded vessels Coronary Artery Disease Reporting and Data System (CAD RADS 5) will be excluded from the study. CCTA is a clinically indicated and standard of care procedure at Lancaster General Hospital.
  .
  Interventions: Device: CT-FFR and CTP

INTERVENTIONS:
Device: CT-FFR and CTP — Those who agree to participate will be scheduled to have the CT-FFR and CTP performed within sixty days of the initial Coronary CTA procedure. A CTA will be performed at rest for FFR. The patient will then take approximately a 30 min break. Regadenoson will then be administered and the dynamic CT procedure will be done for perfusion.

SUMMARY:
This is a prospective, observational study designed to evaluate the role of dynamic computed tomographic perfusion (CTP) and Computed Tomography-Derived Fractional Flow Reserve (CT-FFR) in patients presenting with chest discomfort.Patients with lesions greater than 50% and who meet all other inclusion/exclusion criteria will qualify to be a subject in the CTP study /CT-FFR 49. Those who agree to participate will be scheduled to have the CT-FFR and CTP performed within sixty days of the initial Coronary CTA procedure. A CTA will be performed at rest for FFR. The patient will then take approximately a 30 min break. Regadenoson will then be administered and the dynamic CT procedure will be done for perfusion. If patients are deemed to be appropriate for invasive angiography by the referring physician, coronary lesions between 40% and 80% will get a fractional flow measurement performed if indicated on a clinical basis. Stenosis in vessels less than 1.5 mm will be excluded from the study. The CT-FFR and CTP will be performed in these patients within 60 days of index coronary angiography.

DETAILED DESCRIPTION:
Coronary artery computed tomographic angiography (CCTA) is a widely used, highly accurate technique for the detection of coronary artery disease (CAD), with sensitivity and negative predictive values of over 90% 1-4. Patients with normal CCTA findings have an excellent prognosis and do not require further testing for CAD 5. However, like invasive coronary angiography (CATH), CCTA is an anatomic test and, cannot reliably predict the impairment of flow (functional significance) of Coronary stenoses.

For this reason, in approximately 15-25% of patients, additional functional testing may be required after CCTA, usually in the form of stress testing 6-8. Stress testing is commonly done by exercise or pharmacologic stress with electrocardiographic monitoring and often, imaging of myocardial perfusion by nuclear scintigraphy (MPI) or detection of abnormal contraction by echocardiography. Furthermore, in patients with previously known CAD, CCTA alone is not an adequate test, because in most cases there are multiple lesions that are possible sources of ischemia. Over the last two decades the number of abnormal stress studies have decreased substantially from 40.9% in 1991 to 8.7% in 20099. This underscores the need for an accurate mechanism to identify which patients best benefit from invasive angiography.

Myocardial Computed Tomographic Perfusion (CTP) and Computed Tomography-Derived Fractional Flow Reserve (CT-FFR) have emerged as promising ways to identify ischemia when there is coronary disease identified by CCTA. The two tests provide different and perhaps complimentary information. Fractional Flow Reserve (FFR) measures the difference in flow created by a coronary stenosis before and after the administration of a vasodilator agent by measuring the drop in pressure across the stenosis. Coronary Flow Reserve (CFR) measures flow at maximum vasodilation versus flow at rest in a given arterial tree.

This is a prospective, observational study designed to evaluate the role of dynamic computed tomographic perfusion (CTP) and Computed Tomography-Derived Fractional Flow Reserve (CT-FFR) in patients presenting with chest discomfort.Patients with lesions greater than 50% will qualify to be a subject in the CTP study /CT-FFR 49. Those who agree to participate will be scheduled to have the CT-FFR and CTP performed within sixty days of the initial Coronary CTA procedure. A CTA will be performed at rest for FFR. The patient will then take approximately a 30 min break. Regadenoson will then be administered and the dynamic CT procedure will be done for perfusion. If patients are deemed to be appropriate for invasive angiography by the referring physician, coronary lesions between 40% and 80% will get a fractional flow measurement performed if indicated on a clinical basis. Stenosis in vessels less than 1.5 mm will be excluded from the study. The CT-FFR and CTP will be performed in these patients within 60 days of index coronary angiography.

The CT scanner to be used for this study is an Aquilion ONE ViSION edition 320-detector row scanner with 0.5-mm nominal width detector elements (Toshiba Medical Systems, Otawara, Japan). The scanner has a minimum rotation time of 275 ms. The CT acquisition software includes a novel dose reduction technology (Adaptive Iterative Dose Reduction 3D (AIDR 3D) Toshiba Medical Systems, Otawara, Japan).

Prior to imaging procedures

Patients will have two 18-20 gauge intravenous lines placed, one preferably in an anticubital vein for contrast administration.

Coronary CTA for FFR

All patients receive sublingual nitroglycerine prior to scanning to ensure coronary vasodilatation, while additional oral and/or intravenous beta-blockers will be administered to achieve a pre-scan heart rate of <75 beats per minute (bpm).

For CT-FFR, a standard protocol for coronary CTA will be applied, according to the established protocol at Lancaster General Hospital. Prior to the scan, an automated bolus tracking algorithm (SUREStart) will be used to time the image acquisition to occur during the arterial phase at or near peak contrast. Scan parameters will be as follows: single heart beat half-scan volume acquisition mode with detector collimation 320 x 0.5 mm or less as necessary to cover heart (typically 120 mm); tube voltage 100-120 kV; gantry rotation time 270 ms. To adjust for patient size, tube potential (kV) and tube current (mA) are determined with use of automatic exposure control (SUREExposure3D, and SUREkV, Toshiba Medical Systems). These features reduce variances in image quality by adjusting the acquisition parameters for body habitus.

Prospective electrocardiogram (ECG) triggering will be used to obtain 70-99% of the R-R interval. Radiation dose relevant indices (CT dose index (CTDI vol), dose length product (DLP), and patient size) will be obtained for each examination. Size Specific Dose Estimates (SSD) and Effective Dose (ED) will be calculated by using conversion factors according to standard methodology.

Four phases of the R-R Interval (RR) will be reconstructed covering the range from 70% - 99% (typically 70%, 80%, 90%, and 99%). Reconstruction parameters will be as follows: Medium Calibrated Field of View (CFOV), Filter Convolution (FC) 03 reconstruction kernel, 0.5 mm acquisition thickness with 0.25mm interval, AIDR 3D iterative reconstruction. Adaptive motion correction and FIRST will be used if available.

Dynamic CTP procedure

The CTP procedure involves infusion of a stress agent and a contrast bolus prior to image acquisition. See Figure 2 for a representation of the CTP procedure, and Table 1 for CTP parameters.

No stress agent is FDA-approved specifically for use in CT perfusion. The investigator's choice of stress agent for this study is regadenoson (Lexiscan), a vasodilator widely used in standard-of-care nuclear stress testing. It has been used previously in CT perfusion (12). Regadenoson was chosen for its ease of use and its favorable safety/tolerability profile in patients (37). Its mechanism of action is vasodilation of the coronary vasculature and augmentation of coronary blood flow. Arteries with hemodynamically significant stenosis are not as capable of augmenting flow, resulting in relative under-perfusion in the downstream territory.

The invesitgators will use the standard intravenous dose of Lexiscan recommended for use in nuclear stress testing in this population, which is 5 ml (0.4 mg). Lexiscan, which comes in a prefilled 5 ml syringe containing 0.4 mg of regadenoson, is administered as a rapid (approximately 10-15 seconds) injection into a peripheral vein followed immediately by a 5 ml saline flush. Addendum 1 gives detailed study procedures for myocardial CT perfusion, including the use of Lexiscan, and Addendum 2 gives the Lancaster General Hospital Lexiscan Administration Guidelines.

A 12 lead ECG will be performed at baseline. After this, rhythm monitor leads for CT will be placed. Patient will be positioned supine on the on the CT gantry with continuous ECG monitoring after the baseline ECG is performed as above. If heart rate is greater than 65 beats/minute and blood pressure is greater than 100/60 mm of mercury metoprolol will be administered as per established Lancaster General Health (LGH) protocol for Coronary CTA. Regadenoson will be injected at 0.4 mg / ml followed by 5 ml saline Flush. One minute after regadenoson administration the scanner will be instructed to acquire the heart rate and adjust the gantry rotation time. If patients is stable and has a steady heart rate, 50 cc of contrast will be administered no later than 1.5 minutes after the administration of regadenoson followed by 30 cc - 50 cc of normal saline. The rate of injection for both contrast and saline is 6m/s. A prospectively gated scan will be performed at 70% - 80% of the R - R cycle for every heart beat for a total of 25 seconds. Myocardial Blood flow will be calculated for 17 segments (Table I) . A 12 lead ECG will be obtained immediately after acquisition of images and each subsequent minute for 5 minutes. In the event of ECG changes, the ECG will be repeated every 60 to 90 seconds until it returns to baseline.

For patients who experience stress induced adverse reactions during CTP, aminophylline will be administered IV by a co-investigator physician at a dose of 50-250 mg, using the lowest effective dose. Intravenous Aminophylline is a non-selective phosphodiesterase inhibitor that is FDA approved for the treatment of symptoms and reversible airway obstruction due to asthma and other chronic lung diseases. In addition, it is widely accepted as the primary reversal agent of adenosine, dipyridamole, and regadenoson when patients experience pharmacologic vasodilator stress induced adverse reactions during nuclear cardiac stress testing. The dose used for reactions during stress testing, and which the investigator will use for reactions during CTP, is lower than the FDA approved dose of 5.7 mg/kg dose used in patients with acute symptoms of lung disease.

The CTP examination will be graded using the standard 17-segment myocardial model recommended by the American College of Cardiology Foundation / American Heart Association for nuclear myocardial perfusion and stress echocardiography, in comparison to the myocardial appearance from the baseline coronary CTA. Areas of myocardial hypo-enhancement (decreased CT signal) under hyperemic conditions (coronary vasodilation during the regadenoson infusion) indicate possible ischemia.

Clinical follow-up

If clinically indicated by the initial CCTA and the study CTP, the invasive angiography will be performed at the discretion of the evaluating cardiologist based on a clinical evaluation. Lesions between 40% and 80% will have an FFR. Patients' coronary angiography and FFR will be as per the protocol in Penn Medicine Lancaster General Health.

Long Term Follow-up

Patients medical charts will be reviewed for long term cardiac related outcomes (MACE events, etc) 1 year after the study procedure. This will not require direct participation from the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Age 45 - 85 years.
2. Clinically indicated coronary CTA with one or more lesions greater than 50% in the epicardial vessels.
3. Referring physician agreement to approach the patient for consent.
4. Informed consent from the patient or authorized representative.
5. Scheduled CTA for CT-FFR and CTP within 60 days of the clinically indicated CCTA and prior to any indicated coronary angiography.

   -

Exclusion Criteria:

1. CCTA complication. After an observation period of at least 20 minutes after the index CCTA, any evidence of MACE, allergy, or any other untoward clinical event that reduces CTP safety or suitability (as defined by attending physician) will exclude a patient from eligibility.
2. Medical record of acute ischemia as evidenced on ECG or positive cardiac biomarkers in the interim between index CCTA and CTA for CT-FFR and CTP. Electrocardiographic evidence of acute ischemia includes acute STEMI (ST elevation equal to or greater than 1mm in two or more leads), ST segment depression and/or T wave inversion (not known to be old and thought to be evidence of ongoing ischemia). Positive cardiac biomarkers include elevated troponin, myoglobin).
3. History of asthma or chronic obstructive pulmonary disease requiring bronchodilators or steroid therapy within the past 3 months.
4. Inability to tolerate beta blockers.
5. Atrio-ventricular block (Type II-III), prolonged QT interval or sick sinus syndrome.
6. Renal insufficiency (creatinine ≥1.6 and/or, Glomerular Filtration Rate (GFR) < 60 ml/m) or renal failure requiring dialysis
7. Atrial fibrillation or other markedly irregular rhythm.
8. Psychological unsuitability or extreme claustrophobia.
9. BMI > 35.
10. Pregnancy or unknown pregnancy status.
11. Clinical instability as deemed by the attending physician; including but not limited to: cardiogenic shock, hypotension (systolic blood pressure < 90 mmHg), refractory hypertension (systolic blood pressure > 180 mmHg), sustained ventricular or atrial arrhythmia requiring intravenous medications.
12. Use of Viagra or Cialis in the past 24 hours.
13. Known history of allergy or adverse reactions to x-ray dye, regadenoson or aminophylline.
14. Use of caffeine within the previous 12 hours (inactivates regadenoson).
15. History of severe aortic stenosis.
16. Left main disease greater than 50% and occluded vessels (CAD RADS 5) identified by index Coronary CTA
17. Left Ventricular Ejection Fraction (LVEF) of less than 30%.
18. Significant radiation exposure in the past 18 months (>5 rems OR 2 nuclear or CT studies)
19. Contraindication to CT-FFR: History of myocardial infarction (MI), chronic total occlusions (CTO), stent insertion or PCI, coronary artery bypass grafting (CABG), or arrhythmias; presence of anomalous coronary arteries, anomalous origins of the coronary arteries, or a single coronary artery.

    -

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll patients who have chest discomfort and will require further evaluation for the presence of coronary artery disease. Patients in the study will include those who have had a clinically indicated CCTA for suspicion of coronary artery disease and are determined to have a coronary stenosis ≥50% and ≤99%. However, patients with Left main disease greater than 50% and occluded vessels (CAD RADS 5) will be excluded from the study. CCTA is a clinically indicated and standard of care procedure at Lancaster General Hospital. See Figure 2 for CT Perfusion Workflows at Lancaster General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
Performance of dynamic CTP and CT-FFR for each vessel assessed in patients presenting with chest pain. | Day of imaging (processing of CT-FFR images and reading of CTP images expected to be performed within 48 hours of imaging)
  Performance of CT-FFR compared to CTP for each vessel assessed, as per the below common suite of measures: sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), accuracy, discrimination

SECONDARY OUTCOMES:
Cardiac Long Term Outcomes | MACE: One year from imaging; Performance compared to invasive FFR: Day of imaging for CT-FFR and CTP, invasive FFR performed within 60 days of imaging; Agreement in imaging subsets: Day of imaging
  One-year incidence of MACE events for subjects that undergo CTP and CT-FFR.
Compare measures of CTP and CT-FFR with Coronary Angiography and invasive FFR (in cases where clinically indicated) | MACE: One year from imaging; Performance compared to invasive FFR: Day of imaging for CT-FFR and CTP, invasive FFR performed within 60 days of imaging; Agreement in imaging subsets: Day of imaging
  Sensitivity, specificity, PPV, NPV, accuracy, and discrimination of CTP and CT-FFR compared to invasive FFR. Invasive FFR results may be obtained during Coronary Angiography in cases where clinically indicated. If FFR is not performed by invasive angiography a reference standard of >50% stenosis by invasive coronary angiography will be taken when conventional stress testing has demonstrated ischemia in the distribution supplied by the vessel with stenosis.
Outcome agreement CTP and CT-FFR (when CT-FFR values are <.80 and >0.80 | MACE: One year from imaging; Performance compared to invasive FFR: Day of imaging for CT-FFR and CTP, invasive FFR performed within 60 days of imaging; Agreement in imaging subsets: Day of imaging
  Agreement between CTP and CT-FFR when CT-FFR values are < .80 and >0.80.

CONTACTS AND LOCATIONS:
Overall Officials: Ron M Jacob, MD, Principal Investigator — Penn Medicine/Lancaster General Health
Locations (1):
- Penn Medicine / Lancaster General Hospital, Lancaster, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Budoff MJ, Dowe D, Jollis JG, Gitter M, Sutherland J, Halamert E, Scherer M, Bellinger R, Martin A, Benton R, Delago A, Min JK. Diagnostic performance of 64-multidetector row coronary computed tomographic angiography for evaluation of coronary artery stenosis in individuals without known coronary artery disease: results from the prospective multicenter ACCURACY (Assessment by Coronary Computed Tomographic Angiography of Individuals Undergoing Invasive Coronary Angiography) trial. J Am Coll Cardiol. 2008 Nov 18;52(21):1724-32. doi: 10.1016/j.jacc.2008.07.031. PMID 19007693
- [Background] Hamon M, Biondi-Zoccai GG, Malagutti P, Agostoni P, Morello R, Valgimigli M, Hamon M. Diagnostic performance of multislice spiral computed tomography of coronary arteries as compared with conventional invasive coronary angiography: a meta-analysis. J Am Coll Cardiol. 2006 Nov 7;48(9):1896-910. doi: 10.1016/j.jacc.2006.08.028. Epub 2006 Sep 26. PMID 17084268
- [Background] Meijboom WB, Meijs MF, Schuijf JD, Cramer MJ, Mollet NR, van Mieghem CA, Nieman K, van Werkhoven JM, Pundziute G, Weustink AC, de Vos AM, Pugliese F, Rensing B, Jukema JW, Bax JJ, Prokop M, Doevendans PA, Hunink MG, Krestin GP, de Feyter PJ. Diagnostic accuracy of 64-slice computed tomography coronary angiography: a prospective, multicenter, multivendor study. J Am Coll Cardiol. 2008 Dec 16;52(25):2135-44. doi: 10.1016/j.jacc.2008.08.058. PMID 19095130
- [Background] Miller JM, Rochitte CE, Dewey M, Arbab-Zadeh A, Niinuma H, Gottlieb I, Paul N, Clouse ME, Shapiro EP, Hoe J, Lardo AC, Bush DE, de Roos A, Cox C, Brinker J, Lima JA. Diagnostic performance of coronary angiography by 64-row CT. N Engl J Med. 2008 Nov 27;359(22):2324-36. doi: 10.1056/NEJMoa0806576. PMID 19038879
- [Background] Abdulla J, Asferg C, Kofoed KF. Prognostic value of absence or presence of coronary artery disease determined by 64-slice computed tomography coronary angiography a systematic review and meta-analysis. Int J Cardiovasc Imaging. 2011 Mar;27(3):413-20. doi: 10.1007/s10554-010-9652-x. Epub 2010 Jun 12. PMID 20549366